CLINICAL TRIAL: NCT06778408
Title: Hybrid Arc Palliative Radiation Therapy (HART): A Single Arm Phase II Trial
Acronym: HART
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Vermont Medical Center (Other)
Responsible Party: Principal Investigator, Nataniel Lester-Coll, Assistant Professor, University of Vermont Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UVMC2407/STUDY00003447
Record Dates: First submitted 2025-01-10; First posted 2025-01-16 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Palliative Radiotherapy; Metastatic Cancer (Different Solid Tumour Types)
Keywords: palliative; radiotherapy
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hybrid Arc Palliative Radiation Therapy (Experimental): All patients will receive Hybrid Palliative Radiation Therapy.
  Interventions: Radiation: Hybrid Palliative Radiation Therapy

INTERVENTIONS:
Radiation: Hybrid Palliative Radiation Therapy — Hybrid Palliative Radiation Therapy will be administered to all patients.

SUMMARY:
This is a prospective single-center single-arm Phase II trial of HART for patients with metastatic cancer. The primary objective is to assess the incidence of acute GI toxicity following HART. PRO-CTCAE GI scores observed in the study patients will be compared to historical rates. Secondary outcomes include measuring changes in health-related quality of life, esophageal quality of life, toxicity, dosimetric outcomes, and pain.

DETAILED DESCRIPTION:
Palliative radiation therapy is often used to improve quality of life for patients with metastatic cancer, but severe gastrointestinal (GI) toxicities can limit its effectiveness. HART (Hybrid Arc Radiation Therapy) combines dynamic conformal arcs with conventional radiation beams to deliver more precise dose distributions while sparing healthy organs. This study explores whether HART can reduce acute GI toxicities compared to traditional methods, using validated measures like PRO-CTCAE scores. The goal is to improve patient adherence, reduce side effects, and enhance quality of life, while addressing the lack of clinical data on HART's safety and effectiveness in palliative care.

ELIGIBILITY:
Inclusion Criteria:

Histological confirmation of cancer with radiographic (CT, MRI or PET) evidence of metastatic disease

Palliative radiotherapy indicated for bone or soft tissue metastases, or primary targets, located in the thorax, abdomen, or pelvis as part of their standard of care treatment plan

Age ≥ 18 years.

Women of child-bearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

In lieu of a pregnancy test, participants may sign the Pregnancy Attestation Form, a standard form routinely used in clinical practice at UVMCC.

Recommended methods of birth control are:

The consistent use of an approved hormonal contraception (birth control pill/patches, rings), An intrauterine device (IUD), Contraceptive injection (Depo-Provera), Double barrier methods (Diaphragm with spermicidal gel or condoms with contraceptive foam), Sexual abstinence (no sexual intercourse) or Sterilization.

Men must agree to use a condom and not father a child or donate sperm for the duration of the study and for 90 days after completion of therapy.

A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

* Has not undergone a hysterectomy or bilateral oophorectomy; or
* Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).

Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

Patients receiving any other investigational agents or concurrent cytotoxic chemotherapy

Patients who are pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.

Serious medical comorbidities, which in the opinion of the radiation oncologist preclude the delivery of RT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute gastrointestinal (GI) toxicity | 4 weeks
  Th incidence of acute gastrointestinal (GI) toxicity (defined as a score of ≥2) at 4 weeks post-treatment initiation will be measured and compared to historical data, using PRO-CTCAE GI scores to determine if HART reduces GI toxicity.

SECONDARY OUTCOMES:
patient-reported health-related quality of life | 4 weeks
  Changes in patient-reported health-related quality of life (HRQOL) following HART treatment will be measured, as assessed by the EORTC QLQ-C15-PAL questionnaire from baseline measurements.
patient-reported esophageal quality of life | 4 weeks
  To assess changes in patient-reported esophageal quality of life (QOL) following HART, as measured by the Esophageal Cancer Subscale (ECS) of the FACT-E for thoracic disease, from baseline measurements.
physician graded toxicity | 4 weeks
  Assess physician graded toxicity using NCI-CTCAE v5.
dosimetric outcomes of HART | 4 weeks
  To compare the dosimetric outcomes of HART and conventional AP/PA plans by analyzing dose-volume histograms, with a specific focus on the gastrointestinal organs at risk.
pain scale | 4 weeks
  To evaluate pain scale changes as a surrogate marker for tumor response from baseline to post-HART.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No
Anonymized patient related data will be incorporated into publications and will be made available to other investigators at reasonable request.